CLINICAL TRIAL: NCT00231842
Title: A Pilot Phase II Trial of Adjuvant Radiation Therapy "Sandwiched" Between Ifosfamide in Patients With Mixed Mesodermal Tumors
Brief Title: Adjuvant Radiation Therapy With Ifosfamide in Patients With Mixed Mesodermal Tumors of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Mark H. Einstein, Director, Clinical Research for Women's Health, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-02-040
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Uterine Cancer
Keywords: Mixed Mesodermal Tumor; MMT; Uterine Cancer; Radiation Therapy; Chemotherapy
MeSH Terms: conditions — Uterine Neoplasms; Mixed Tumor, Mesodermal | interventions — Ifosfamide; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Ifosfamide with or without cisplatin (Experimental): Participants with surgically staged carcinosarcoma (CS) with no gross residual disease were initially administered ifosfamide (1.2 g/m2/day for 5 days) with cisplatin (20 mg/m2/day for 5 days) every 3 weeks for 3 cycles followed by pelvic external beam RT and brachytherapy followed by 3 additional cycles of ifosfamide (1.0 g/m2/day) with cisplatin with cisplatin (20 mg/m2/day for 5 days) evrey 3 weeks. cisplatin added toxicity without additional efficacy, so mid-study, cisplatin was eliminated.
  Interventions: Drug: Ifosfamide; Device: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Ifosfamide — Ifosfamide 1.2gm/m2/day for 5 days. Mesna 400mg/IV bolus at each ifosfamide dosing followed by 1200mg IV divided in 3L / day x 5 days. Repeat q21 days x 3 cycles. After 3 cycles, RT. After RT, Ifosfamide 1.0gm/m2/day for 5 days. Mesna 333 mg/IV bolus at each ifosfamide dosing followed by 1000mg IV divided in 3L /day x 5 days. Repeat q21 days x 3 cycles.
Device: Radiation Therapy — Ifosfamide 1.2gm/m2/day for 5 days. Mesna 400mg/IV bolus at each ifosfamide dosing followed by 1200mg IV divided in 3L / day x 5 days. Repeat q21 days x 3 cycles. After 3 cycles, RT. After RT, Ifosfamide 1.0gm/m2/day for 5 days. Mesna 333 mg /IV bolus at each ifosfamide dosing followed by 1000mg IV divided in 3L /day x 5 days. Repeat q21 days x 3 cycles.
  Other Names: Pelvic RT, Radiation
Drug: Cisplatin — dosage is 20 mg/m2/day for 5 days, ever 3 weeks.

SUMMARY:
The optimal sequence and /or modality for adjuvant therapy in the management of Mixed Mesodermal Tumors (MMT) clearly remains to be established. The rationale for the protocol is to "sandwich" pelvic radiation with chemotherapy to decrease distant metastasis.

The proposed study will sandwich radiation between the two most active chemotherapeutic agents for MMT identified to date (ifosfamide/cisplatin). By doing so, we attempt to decrease both local and distant recurrence, which may translate into an improved progression free interval and possibly even extend survival.

DETAILED DESCRIPTION:
Uterine sarcomas account for only 2-4% of uterine malignancies, yet they are responsible for 26% of uterine cancer deaths. Mixed mesodermal tumors (MMT), previously known as carcinosarcoma, are the most common of the uterine sarcomas in the United States. Prognosis for these patients is generally grim due to the propensity for early metastatic disease. Patterns of spread are by both hematogenous and lymphatic dissemination. It has been noted that 66% of patients with disease clinically confined to the uterus have nodal metastasis at the time of diagnosis. The majority of patients will die with both wide spread intra-abdominal and pelvic disease within two years of diagnosis.

Adjuvant pelvic radiation therapy has been advantageous in controlling local recurrence. One study reports 26% local recurrence in patients treated with surgery alone versus 14% recurrence in patients treated with surgery and adjuvant pelvic radiation. Although adjuvant radiation shows a benefit in improving local control, it has not been found to impact survival. This finding is likely attributed to the high incidence of distant metastasis (85%) known to occur with disease recurrence.

Multiple chemotherapeutic agents have been evaluated in the management of advanced, persistent or recurrent uterine MMT. Response to single agent therapy has been less than 35% with the most active agents identified being ifosfamide (response rate = 34.8%) and cisplatin (response rate 17.9%. The use of chemotherapy in the adjuvant setting has been explored as a means of attempting to impact the incidence of distant metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented mixed mesodermal tumor (MMT) of uterus with no visible residual disease.
* Surgical staging to include total abdominal hysterectomy, bilateral salpingo-oophorectomy, peritoneal washings, and lymph node sampling.
* Surgical staging should be completed 6 weeks ± 7 days prior to enrollment.
* Age >= 18 years.
* Written voluntary informed consent.

Exclusion Criteria:

* Patient has impairment of hepatic, renal or hematologic function as defined by the following baseline laboratory values:

  * Total serum bilirubin >1.5mg/dl
  * History of chronic or active hepatitis
  * Serum creatinine >2.0 mg/dl
  * Platelets <100,000/mm3
  * Absolute neutrophil count (ANC) <1500/mm3
  * Hemoglobin <8.0 g/dl (the patient may be transfused prior to study entry)
* Patient has severe or uncontrolled medical disease (eg. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.)
* Patient has been treated with myelosuppressive chemotherapy within three weeks prior to study entry.
* Patients with any prior chemotherapy or radiotherapy for pelvic malignancy.
* Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at time of study entry.
* Patient has a uterine sarcoma other then mixed mesodermal tumor (MMT).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Einstein, M.D., M.S., Principal Investigator — Montefiore Medical Center and Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Einstein MH, Klobocista M, Hou JY, Lee S, Mutyala S, Mehta K, Reimers LL, Kuo DY, Huang GS, Goldberg GL. Phase II trial of adjuvant pelvic radiation "sandwiched" between ifosfamide or ifosfamide plus cisplatin in women with uterine carcinosarcoma. Gynecol Oncol. 2012 Jan;124(1):26-30. doi: 10.1016/j.ygyno.2011.10.008. Epub 2011 Nov 3. PMID 22055846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants with surgically staged I-IV uterine carcinosarcoma (CS) without evidence of gross residual disease after primary surgery were recruited from 1999 to 2009 . Eligible participants underwent surgical staging when clinically indicated.
Pre-assignment Details: 30 participants were enrolled and 3 participants withdrew prior to therapy. Twenty-seven participants received the first three cycles of chemotherapy and Radiation Therapy and were included in the analysis.
Groups:
- Chemotherapy and Radiation Therapy: Participants with surgically staged carcinosarcoma (CS) with no gross residual disease were initially administered ifosfamide (1.2 g/m2/day for 5 days) with cisplatin (20 mg/m2/day for 5 days) every 3 weeks for 3 cycles followed by pelvic external beam RT and brachytherapy followed by 3 additional cycles of ifosfamide (1.0 g/m2/day) with cisplatin with cisplatin (20 mg/m2/day for 5 days) evrey 3 weeks. cisplatin added toxicity without additional efficacy, so mid-study, cisplatin was eliminated.
Period: Overall Study
Arm/Group | Chemotherapy and Radiation Therapy
Started | 30
Initiated Therapy | 27
Completed First 3 Cycles (27 participants completed the first 3 cycles of chemotherapy followed by RT) | 27
Completed Prescribed RT (26 participants had EBRT + Brachytherapy; 1 had EBRT alone) | 27
Completed Full Prescribed Therapy | 19
Completed | 19
Not Completed | 11
Not completed — Withdrawal by Subject | 3
Not completed — Did not complete the last 3 cycle | 8

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy and Radiation Therapy: Adjuvant Radiation Therapy "Sandwiched" between Ifosfamide in Patients with Mixed Mesodermal Tumors
  Radiation Therapy : Ifosfamide 1.2gm/m2/day for 5 days. Mesna 400mg/IVSS bolus at each ifosfamide dosing followed by 1200mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles. After 3 cycles, RT. After RT, Ifosfamide 1.0gm/m2/day for 5 days. Mesna 333mg/IVSS bolus at each ifosfamide dosing followed by 1000mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles.
  Ifosfamide : Ifosfamide 1.2gm/m2/day for 5 days. Mesna 400mg/IVSS bolus at each ifosfamide dosing followed by 1200mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles. After 3 cycles, RT. After RT, Ifosfamide 1.0gm/m2/day for 5 days. Mesna 333mg/IVSS bolus at each ifosfamide dosing followed by 1000mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles.
Arm/Group | Chemotherapy and Radiation Therapy
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27
FIGO Staging [Count of Participants; unit: Participants] — Federation of Gynecology and Obstetrics (FIGO) is a system for staging gynecologic cancer.
  I Malignancy of one (Ia) or both (Ib) ovaries, without ascites; 5-year survival: 60%
  II Malignancy of one (IIa) or both (IIb) ovaries, with pelvic extension and ascites; 5-year survival: 40%
  III Malignancy involves one/both ovaries, intraperitoneal metastases outside pelvis and/or positive retroperitoneal lymph nodes; 5-year survival: 5%
  IV Involvement of one/both ovaries with metastases and histologically confirmed extension to pleural cavity or liver; 5-year survival, 3%
  Participants
    Total Stage I | 14
    Total Stage II | 3
    Total Stage III | 7
    Total Stage IV | 3

OUTCOME MEASURES:

1. Primary Outcome: Cycles With Hematologic Toxicities
Description: Out of 162 planned cycles, a total of 138 cycles (85%) were administered. Number of cycles during which participants with grades 3 and 4 experienced hematologic toxicities are reported. Most of the toxicities were self-limiting.
Time Frame: 2 years
Measure: Number; unit: Cycles
Groups:
- Grade 3 Toxicity: Adjuvant Radiation Therapy "Sandwiched" between Ifosfamide in Patients with Mixed Mesodermal Tumors
  Ifosfamide: Ifosfamide 1.2gm/m2/day for 5 days. Mesna 400mg/IVSS bolus at each ifosfamide dosing followed by 1200mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles. After 3 cycles, RT. After RT, Ifosfamide 1.0gm/m2/day for 5 days. Mesna 333mg/IVSS bolus at each ifosfamide dosing followed by 1000mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles.
  Radiation Therapy: Ifosfamide 1.2gm/m2/day for 5 days. Mesna 400mg/IVSS bolus at each ifosfamide dosing followed by 1200mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles. After 3 cycles, RT. After RT, Ifosfamide 1.0gm/m2/day for 5 days. Mesna 333mg/IVSS bolus at each ifosfamide dosing followed by 1000mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles.
- Grade 4 Toxicity: Adjuvant Radiation Therapy "Sandwiched" between Ifosfamide in Patients with Mixed Mesodermal Tumors
  Ifosfamide: Ifosfamide 1.2gm/m2/day for 5 days. Mesna 400mg/IVSS bolus at each ifosfamide dosing followed by 1200mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles. After 3 cycles, RT. After RT, Ifosfamide 1.0gm/m2/day for 5 days. Mesna 333mg/IVSS bolus at each ifosfamide dosing followed by 1000mg IV divided in 3L/day x 5 days. Repeat q21 days x 3 cycles.
Arm/Group | Grade 3 Toxicity | Grade 4 Toxicity
Number analyzed (Participants) | 27 | 27
Cycles
  Neutropenia | 11 | 14
  Anemia | 6 | 0
  Thrombocytopenia | 6 | 2

ADVERSE EVENTS:
Time Frame: Participants were followed up to 2 years.
Description: Adverse events were monitored for each cycle during therapy and during follow-up and graded using the National Cancer Institute Common Toxicity Criteria (CTC) version 3.0. Frequencies for toxicity and adverse events were recorded.
  Although adverse events were monitored, however, not all adverse events are being reported. The PI and the study team have left the institution. Sincere efforts were made to obtain the data, however, the adverse events data is not available.
Arm/Group | Chemotherapy and Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 13/27
Other Adverse Events (participants affected / at risk) | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy and Radiation Therapy (N=27)
Neutropenia (Blood and lymphatic system disorders) | 13 — low count of white blood cells.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No